CLINICAL TRIAL: NCT03369678
Title: Promoting Health Equity for Indigenous and Non-Indigenous People in Emergency Departments
Brief Title: EQUIP Emergency: Promoting Health Equity for Indigenous and Non-Indigenous People in Emergency Departments
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Colleen Varcoe, Professor, University of British Columbia
Other Study IDs: H17-01548
Record Dates: First submitted 2017-11-18; First posted 2017-12-12 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Interventions to Enhance Emergency Health Care
Keywords: Cultural Safety; Discrimination; Emergency Departments; Health Equity; Indigenous Populations; Marginalized Populations; Patient Experiences of Care; Trauma- and Violence-Informed Care; Staff Engagement; Harm Reduction
MeSH Terms: conditions — Emergencies; Wounds and Injuries; Harm Reduction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emergency Departments (EDs) in Canada often operate over-capacity and are under significant pressures. In this environment, particular groups of people experience inadequate and inequitable treatment in EDs, including Indigenous people, racialized newcomers, people with mental illnesses, those living in unstable housing or facing homelessness, experiencing interpersonal violence or using substances, and people involved in sex work. Stigma and discrimination in health care deter people from accessing care, interfering with effective care delivery, increasing reliance on EDs, and increasing human and financial costs. This project will develop and test a framework for health equity interventions to promote the provision of equity-oriented care in EDs.

DETAILED DESCRIPTION:
This study examines the feasibility, process, and impacts of implementing an evidence-informed framework for interventions to enhance the capacity of Emergency Departments to provide high-quality care to people at greatest risk of experiencing health and health care inequities. The framework integrates evidence-based strategies to mitigate discrimination and racism experienced by Indigenous people, and stigma and discrimination faced by people of all ethnicities related to substance use, housing instability, sex work, gender, or mental illnesses. The study tests organizational interventions that incorporate principles of equity-oriented care, trauma- and violence-informed care, harm reduction, and cultural safety to optimize care first for Indigenous people, and then for a range of people who commonly face stigma and discrimination.

Approaching EDs as complex adaptive systems, the study aims to:

1. Engage EDs in a participatory process to enhance capacity for equity-oriented care
2. Examine impacts of equity-oriented interventions on processes of care, patient experiences of care and short-term outcomes, staff attitudes, confidence, behaviours and job satisfaction, and cost
3. Analyze the cost-effectiveness and feasibility of implementing the interventions and scale-up potential in other contexts.

This mixed-methods study incorporates administrative data, survey data with standardized tools, in-depth interviews, analysis of policy and organizational structures, and observational data. The study is divided into multiple phases of data collection. This phase focuses on surveys of ED staff members and patients. The structured surveys use standardized tools and measures, and aim to capture staff and patients' experiences of ED care. Surveys will be conducted at three to four timepoints.

PATIENT SURVEYS will draw on patient self-reports to measure changes over time in processes of care and perceived quality of care. These indicators will be measured through structured, researcher-facilitated surveys conducted with a sample of 250-300 patients at each site at up to four points in time, providing pre- and post-intervention comparisons.

At each data collection point, all patients who are able to provide informed consent (in the languages available - see below) will be invited to participate as they present for care or during the course of their visit at each emergency unit. Researchers will circulate throughout the emergency department, inviting participation by all patients who are conscious and able to consent.

Recruitment will occur over a period of 1-3 weeks in 6 hour blocks. The blocks will span all 24 hours, and as many days of the week as possible.

Surveys will not delay or interrupt provision of care.

Section 1 of the survey can be completed at any time during the patient's Emergency visit; Section 2 will be completed after the patient has been cleared for discharge from the Emergency (discharged to community or admitted). The system for notifying the researchers of discharge status will align with the usual procedures at each ED. If at all possible, Section 2 will be completed before the patient leaves the hospital, in a private space close to the ED. If the patient is unable or prefers not to complete Section 2 in hospital, then a phone follow up will be offered; if the patient does not have a phone and is willing and able to do so, they will be invited to drop in at a specified outpatient or community clinic in the following 5 days.

Recruitment and data collection will continue until target samples of 250-300 completed surveys per site per time point are achieved. Every effort will be made to recruit participation of people from diverse ethnocultural groups. Given the research objectives of this study, recruitment will be prioritized for people who self-identify as Indigenous as well as individuals who are at risk of experiencing stigma and discrimination (e.g., those with diagnoses related to mental illness, HIV, substance use).

Researchers will work in pairs during each time block conducting recruitment and interviewing simultaneously. Following processes already in use at one of the partnering ED sites and prior practices, researchers will collect data directly on tablets using structured survey instruments.

A team of trained researchers will work with ED staff members (e.g., triage staff, unit clerk, charge nurse, etc.), to invite participation by those patients who meet the established eligibility criteria. In urgent cases, participants will be told about the study by staff after their immediate/urgent health concerns have been addressed. Researchers will approach potential participants to explain the study and seek consent to participate. Once consent is obtained, the researcher will enroll the participant in the study, complete Section 1 of the survey, and collect minimal contact information (i.e., name and phone number - see Patient Survey Guide) to be used for follow up in the event that patients elect to be interviewed by phone or off-site at a later time.

The brief structured survey (10-15 minutes per section) will be facilitated by a researcher with patients who consent. Both sections will be completed within a maximum of 5 days of the ED visit in a private area close to the ED, where participants' responses cannot be overheard by others and confidentiality can be maintained, or by phone or at an agreed upon drop-in location within the hospital. Patients will be provided with an honorarium for completing each section of the survey. Transportation and childcare expenses will be reimbursed for those who choose an in-person follow up to complete the survey. A detailed safety protocol, adapted from previous studies, will be used to guide all interactions.

Structured surveys conducted in all waves will be facilitated by a trained researcher, following an established Patient Survey Guide and using a computer-assisted data platform (UBC Survey Tool) on a tablet device. This tablet interface will allow the participant and researcher to view questions and select responses together on the screen.

STAFF SURVEYS All staff members at each partnering ED site will be invited to complete a survey questionnaire, which will include measures aligned with the theoretical principles underlying the equity-oriented framework being tested (i.e., cultural safety, trauma- and violence-informed care, and harm reduction).

Staff members will be invited to complete a structured questionnaire (see Staff Survey Guide), to be administered online or completed on paper. To facilitate this, copies of the survey will be available within each emergency department. In addition, in-person sessions will be held at each emergency department. Light refreshments will be provided and researchers will be on-hand to answer any questions about the study and the survey itself. Participants will be encouraged to attend these sessions on their break or at shift-end, and can choose to complete the surveys independently on paper or directly on a study tablet.

A preamble to the survey will explain the study and include the consent form. Completion of the survey - either online or on paper - will imply consent.

Staff assessments will be conducted at three to four time points, to coincide with milestones in the implementation of the intervention being tested. When possible, staff will be encouraged to complete the survey outside of work hours, during breaks, or at the start or end of their shifts.

ELIGIBILITY:
Inclusion Criteria:

PATIENT SURVEYS

* Age 19 or over, or emancipated youth (16-19 years old)*
* Able to provide informed consent.
* Patient presenting for care at a participating ED site when survey recruitment is being conducted * Patients between age 16 and 19 will only be included if they no longer live with a parent or guardian.

STAFF SURVEYS

* Age 19 or over
* Able to understand, read and write in English
* Staff member or health professional working in a participating ED site

Exclusion Criteria:

* Individuals not meeting the inclusion criteria listed above will be excluded from participation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of three participating emergency departments.
  Staff members of three participating emergency departments.
Sampling Method: Non-Probability Sample
Enrollment: 5439 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patients' overall rating of care post-intervention | Pre-intervention: baseline & 6-9 months; Post-intervention: immediately following intervention period (14-15 months post-baseline #2)
  Change in self-reported rating of care, measured on a scale from 0 to 10, comparing pre-intervention to post-intervention
Change from baseline in patients' overall rating of care at 6-11 months post-intervention | Pre-intervention: baseline & 6-9 months; Post-intervention: 6-11 months after intervention period (21-25 months post-baseline #2)
  Change in self-reported rating of care, measured on a scale from 0 to 10, comparing pre-intervention to post-intervention
Change from baseline in staff perception of patient care post-intervention | Immediately following intervention period (12 months post-baseline)
  Change in staff members' self-reported perception of the patient care provided by their work unit/team, comparing pre-intervention to post-intervention
Change from baseline in staff perception of patient care at 6-12 months post-intervention | 18-25 months post-baseline
  Change in staff members' self-reported perception of the patient care provided by their work unit/team, comparing pre-intervention to post-intervention
Change from baseline in staff perception of patient care at 17 months post-intervention | 29 months post-baseline
  Change in staff members' self-reported perception of the patient care provided by their work unit/team, comparing pre-intervention to post-intervention

SECONDARY OUTCOMES:
Change from baseline in Discrimination in Medical Settings Scale post-intervention | Pre-intervention: baseline & 6-9 months; Post-intervention: immediately following intervention period (at 14 - 15 months post-baseline #2)
  Change in patients' self-reported experiences of discrimination in the emergency department, comparing pre-intervention to post-intervention
Change from baseline in Discrimination in Medical Settings Scale at 6-11 months post-intervention | Pre-intervention: baseline & 6-9 months; Post-intervention: 6-11 months after intervention period (21-25 months post-baseline #2)
  Change in patients' self-reported experiences of discrimination in the emergency department, comparing pre-intervention to post-intervention
Change from baseline in staff satisfaction and engagement post-intervention | Immediately following intervention period (12 months post-baseline)
  Change in staff members' self-reported satisfaction and engagement with their job and workplace, comparing pre-intervention to post-intervention
Change from baseline in staff satisfaction and engagement at 6-12 months post-intervention | 18-25 months post-baseline
  Change in staff members' self-reported satisfaction and engagement with their job and workplace, comparing pre-intervention to post-intervention
Change from baseline in staff satisfaction and engagement at 17 months post-intervention | 29 months post-baseline
  Change in staff members' self-reported satisfaction and engagement with their job and workplace, comparing pre-intervention to post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Varcoe, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - University Hospital of Northern British Columbia, Prince George, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varcoe C, Browne AJ, Perrin N, Wilson E, Bungay V, Byres D, Wathen N, Stones C, Liao C, Price ER. EQUIP emergency: can interventions to reduce racism, discrimination and stigma in EDs improve outcomes? BMC Health Serv Res. 2022 Sep 2;22(1):1113. doi: 10.1186/s12913-022-08475-4. PMID 36050677
- [Derived] Varcoe C, Bungay V, Browne AJ, Wilson E, Wathen CN, Kolar K, Perrin N, Comber S, Blanchet Garneau A, Byres D, Black A, Price ER. EQUIP Emergency: study protocol for an organizational intervention to promote equity in health care. BMC Health Serv Res. 2019 Oct 10;19(1):687. doi: 10.1186/s12913-019-4494-2. PMID 31601199
- See also: EQUIP Health Care website. Click for more info about the EQUIP Emergency study. — https://equiphealthcare.ca/

DOCUMENTS (2):
  • Informed Consent Form: Patient Consent Form (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03369678/ICF_000.pdf
  • Informed Consent Form: Accompanying Person Consent Form (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03369678/ICF_001.pdf